CLINICAL TRIAL: NCT01773200
Title: Prognostic Value of Circulating Endothelial Progenitor Cells in Aneurysmal Subarachnoid Hemorrhage (Evaluation de l'intérêt Pronostic Des progéniteurs endothéliaux Circulants Dans l'hémorragie Sous-arachnoïdienne Par Rupture d'anévrysme cérébral)
Brief Title: Prognostic Value of Circulating Endothelial Progenitor Cells in Aneurysmal Subarachnoid Hemorrhage
Acronym: EVAPROPEC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2012/153
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: endothelial progenitor cells; aneurysmal subarachnoid hemorrhage; vasospasm; BNP
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aneurysmal Subarachnoid Hemorrhage: Each consecutive patient suffering from aneurysmal subarachnoid hemorrhage

SUMMARY:
Aneurysmal subarachnoid hemorrhage is a common and serious disease associated to a high rate of mortality and morbidity. Severe definitive neurological impairment can concern up to 30% of patients in relation with elevated intracranial pressure, hemorrhage recurrence and symptomatic cerebral arterial vasospasm. This latter complication is defined as a reversible reduction of cerebral artery's diameter occurring between the 4th and the 14th day after bleeding. Physiopathology is not well understood, but could involve endothelium, trough endothelial progenitor cells (EPC). Circulating EPC are bone marrow-derived cells with capacity of vasculogenesis and angiogenesis. EPC have been recognized playing a beneficial role in cardiovascular disease and ischemic stroke. EPC have never been studied in aneurysmal subarachnoid hemorrhage.

The primary objective of this study is to compare the number of circulating endothelial progenitor cells between patients with a good neurological outcome (defined as a glasgow outcome scale = 1 or 2) and patients with a poor neurological outcome (glasgow outcome scale = 3, 4 or 5).

Briefly, the number of circulating EPC will be measured at admission, and at day 3, 6, 10, 14, 21 in each consecutive patient suffering aneurysmal subarachnoid hemorrhage and hospitalized in Teaching Hospital of Besançon (France). The neurological outcome will be measured one year after subarachnoid hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* recent(< 24 h) aneurysmal subarachnoid hemorrhage
* written informed consent obtained from the patient or from close relatives

Exclusion Criteria:

* refusal to participate
* Non-aneurysmal subarachnoid hemorrhage
* aneurysmal subarachnoid hemorrhage with estimated date of bleeding > 24 h
* Chronic heart failure
* Chronic medication able to modify the plasmatic level of BNP
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients suffering from acute aneurysmal subarachnoid haemorrhage. .
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2013-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
endothelial progenitor cells count | day 3 after bleeding

SECONDARY OUTCOMES:
Endothelial progenitor cells count | day 0, 6, 10, 14, 21 after bleeding
Maximal amplitude of variation of EPC count | 3 weeks after bleeding
Plasmatic brain natriuretic peptide | day 0, 3, 6, 10, 14, 21 after bleeding

OTHER OUTCOMES:
Glasgow Outcome Scale | One year after bleeding
Vasospasm occurence | during the 3 weeks after bleeding
  Vasospasm will be defined as at less one segmental narrowing of a cerebral artery diagnosed on cerebral angiography (angio scanner, angio-MRI or 4 axes cerebral arteriography). Cerebral angiography will be done as necessary according to the occurence of the following situations
  * a clinical neurological deterioration unexplained by another cause
  * a mean arterial blood flow speed higher than 2 m/s assessed in cerebral arteries by transcranial doppler or a significant elevation of the mean arterial blood flow speed on two consecutive evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Pili-Floury, MD, PhD, Principal Investigator — CHRU de Besançon
Locations (1):
- CHRU de Besançon, Besançon, France